CLINICAL TRIAL: NCT05287958
Title: A Pilot Study on the Technical Feasibility of an Electrical Impedance Tomography Device for Quantitative Pulmonary Function Testing in ALS Patients
Brief Title: Feasibility of an Electrical Impedance Tomography Device for Pulmonary Function Testing in ALS Patients
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Seward Rutkove, Chairman, Department of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2020C-001010; R21NS118434 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-04

CONDITIONS: ALS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy: While no intervention or investigational agent will be used in this study, an EIT system will be used, which is a Non-Significant Risk Device.
  Interventions: Diagnostic Test: EIT
- ALS: While no intervention or investigational agent will be used in this study, an EIT system will be used, which is a Non-Significant Risk Device.
  Interventions: Diagnostic Test: EIT

INTERVENTIONS:
Diagnostic Test: EIT — EIT comprises a chest belt that is connected to a computer via a universal serial bus (USB) or an Ethernet cable. The chest belt captures EIT data, which is transmitted via the USB or Ethernet cable to the computer. Tomography-like impedance images of the lungs are computed and displayed on the computer. The impedance images will be used to evaluate lung recruitment and other pulmonary function parameters that are currently measured using standard-of-care PFT devices.

SUMMARY:
This is an unblinded pilot study to investigate the technical feasibility of using an electrical impedance tomography device for noninvasive pulmonary function monitoring in ALS patients. The study will enroll patients with ALS in one cohort and healthy volunteers in a second cohort that will both undergo EIT imaging with the investigational device prior to and while performing a standard PFT procedure.

DETAILED DESCRIPTION:
This is an unblinded pilot study to investigate the technical feasibility of using an electrical impedance tomography device for noninvasive pulmonary function monitoring in ALS patients.

For both Cohort I and II, subject participation will require two visits (initial and 3-4 month follow up), which are expected to last approximately 30 minutes. Subjects will undergo EIT imaging with the investigational device prior to and while performing a standard PFT procedure. The actual EIT imaging will last for 10 to 15 minutes.

ELIGIBILITY:
Cohort I

Inclusion Criteria:

1. ALS patients able to perform PFT.
2. ALS patients recommended for PFT.
3. Subjects capable of giving written informed consent.
4. Adult, age ≥ 18 years old.

Exclusion Criteria:

1. Serious psychiatric illnesses.
2. Presence of an implanted electronic device (e.g. pacemaker, vagal stimulator, deep brain stimulator) or electrodes or electrical wires.
3. Skin lesions at chest belt placement sites.
4. Pregnant women.
5. Patients with primary lung disease, at the discretion of the Investigator.

Cohort II

1. Subjects capable of giving written informed consent; 2. Subjects capable of performing a PFT; 3. Adult, age ≥ 18 years old 10.2.2 Exclusion Criteria

1. Serious psychiatric illnesses.
2. Presence of an implanted electronic device (e.g. pacemaker, vagal stimulator, deep brain stimulator) or electrodes or electrical wires.
3. Skin lesions at chest belt placement sites.
4. Pregnant women.
5. Subjects with primary lung disease, at the discretion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients clinically diagnosed with ALS
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Correlation of EIT and PFT measures | Through study completion, an average of 3 months
  A correlation coefficient (-1 to +1) will be used

SECONDARY OUTCOMES:
Assessing differences in lung function images in healthy versus ALS cohorts as generated with EIT | Through study completion, an average of 3 months
  Correlation coefficient (-1 to +1) will be used to compare regions of interest

CONTACTS AND LOCATIONS:
Overall Officials: Seward Rutkove, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire